CLINICAL TRIAL: NCT01493531
Title: A Phase 3 Randomized, Double-Blind, Multicenter, Placebo- Controlled, Combination Study to Evaluate the Efficacy and Safety of Lesinurad and Allopurinol Compared to Allopurinol Alone in Subjects With Gout Who Have Had an Inadequate Hypouricemic Response to Standard of Care Allopurinol
Brief Title: Combining Lesinurad With Allopurinol in Inadequate Responders
Acronym: CLEAR 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-302; 2011-003767-29 (EudraCT Number)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lesinurad 200 mg + allopurinol (Experimental)
  Interventions: Drug: Lesinurad; Drug: Allopurinol
- lesinurad 400 mg + allopurinol (Experimental)
  Interventions: Drug: Lesinurad; Drug: Allopurinol
- Placebo + allopurinol (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Allopurinol

INTERVENTIONS:
Drug: Lesinurad — Tablets, 200 mg QD
  Arms: lesinurad 200 mg + allopurinol
Drug: Lesinurad — Tablets, 400 mg QD
  Arms: lesinurad 400 mg + allopurinol
Drug: Placebo — Tablets, Placebo QD
  Arms: Placebo + allopurinol
Drug: Allopurinol — Tablets

SUMMARY:
This study will compare the serum uric acid lowering effects, clinical benefits, and safety of lesinurad in combination with allopurinol to allopurinol alone in subjects with gout who have had an inadequate response to allopurinol.

DETAILED DESCRIPTION:
Allopurinol is the standard of care for the treatment of gout. Nevertheless, most patients treated with allopurinol do not achieve the recommended sUA target of < 6.0 mg/dL and need additional therapy to achieve the target. Probenecid and benzbromarone are URAT1 inhibitors, generally recommended as second-line agents for patients who are either resistant to or intolerant of allopurinol. However, benzbromarone is not available in the US and probenecid is rarely used. Consequently, there is a clear unmet medical need for a new safe and effective therapy for gout, such as lesinurad, a potent URAT1 inhibitor, that can be used in combination with allopurinol in patients not responding adequately to allopurinol monotherapy so that very high rates of response can be achieved by nearly all gout patients, rather than a minority.The subjects selected for this study will have moderate to severe gout with an inadequate response to allopurinol

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject meets the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has been taking allopurinol as the sole urate-lowering therapy indicated for the treatment of gout for at least 8 weeks prior to the Screening Visit at a stable, medically appropriate dose, as determined by the investigator, of at least 300 mg per day (at least 200 mg for subjects with moderate renal impairment).
* Subject must be able to take gout flare prophylaxis with colchicine or an NSAID (including Cox-2 selective NSAID) ±PPI.
* Subject has an sUA level ≥ 6.5 mg/dL at the Screening Visit and ≥ 6.0 mg/dL at Day -7 Visit.
* Subject has reported at least 2 gout flares in the prior 12 months.
* Body mass index (BMI) < 45 kg/m2

Exclusion Criteria:

* Subject with known hypersensitivity or allergy to allopurinol.
* Subject who is taking any other approved urate-lowering medication that is indicated for the treatment of gout other than allopurinol within 8 weeks of the Screening Visit.
* Subject who is pregnant or breastfeeding.
* Subject who consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* Subject with a history or suspicion of drug abuse within the past 5 years.
* Subject that requires or may require systemic immunosuppressive or immunomodulatory treatment.
* Subject with known or suspected human immunodeficiency virus (HIV) infection.
* Subject with a positive test for active hepatitis B or hepatitis C infection.
* Subject with a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer.
* Subject within the last 12 months with: unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis; or subjects currently receiving anticoagulants.
* Subject with uncontrolled hypertension.
* Subject with an estimated creatinine clearance < 30 mL/min.
* Subject with active peptic ulcer disease requiring treatment.
* Subject with a history of xanthinuria, active liver disease, or hepatic dysfunction.
* Subject receiving chronic treatment with more than 325 mg of salicylates per day.
* Subject taking valpromide, progabide, or valproic acid.
* Subject who has received an investigational therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the Screening Visit.
* Subject with any other medical or psychological condition, which might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Ardea Biosciences, Inc.
Locations (158):
- United States (79):
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Pheonix, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Gold River, California
  - Irvine, California
  - La Jolla, California
  - Roseville, California
  - San Diego, California
  - San Ramon, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Glenwood Springs, Colorado
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Brandon, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Plant City, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Dunwoody, Georgia
  - Roswell, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Addison, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Lexington, Kentucky
  - Cumberland, Maryland
  - Wheaton, Maryland
  - Fall River, Massachusetts
  - Hyannis, Massachusetts
  - Ann Arbor, Michigan
  - Flint, Michigan
  - Olive Branch, Mississippi
  - Louis, Missouri
  - Omaha, Nebraska
  - Reno, Nevada
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - Shelby, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Franklin, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Indiana, Pennsylvania
  - Scottdale, Pennsylvania
  - Greenville, South Carolina
  - Greer, South Carolina
  - Spartanburg, South Carolina
  - Union, South Carolina
  - Knoxville, Tennessee
  - Spring Hill, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Irving, Texas
  - Sugarland, Texas
  - West Layton, Utah
  - Danville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Australia (9):
  - Camperdown, New South Wales
  - Wollongong, New South Wales
  - Bisbane, Queensland
  - Herston, Queensland
  - Woodville South, South Australia
  - Clayton, Victoria
  - Heidelberg West, Victoria
  - Perth, Western Australia
  - Shenton Park, Western Australia
- Belgium (6):
  - Genk, Limburg
  - Gozée
  - Kortrijk
  - Lommel
  - Mouscron
  - Yvoir
- Canada (12):
  - Coquitlam, British Columbia
  - Kamloops, British Columbia
  - Penticton, British Columbia
  - Paradise, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Corunna, Ontario
  - Greater Sudbury, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- Germany (9):
  - Kamenz, Saxony
  - Berlin
  - Dresden
  - Eichstätt
  - Goch
  - Leipzig
  - Mannheim
  - Munich
  - Osnabrück
- New Zealand (6):
  - Tauranga, Bay of Plenty
  - Beckenham, Christchurch
  - Garden Place, Hamilton
  - Bay of Plenty, Rotorua
  - Auckland
  - Takapuna
- Poland (10):
  - Krakow, Lesser Poland Voivodeship
  - Bialystok, Podlaskie Voivodeship
  - Elblag, Warmian-Masurian Voivodeship
  - Gmina Końskie
  - Katowice
  - Krakow
  - Poznan
  - Radom
  - Warsaw
  - Wroclaw
- South Africa (17):
  - Fichardtpark, Bloemfontein
  - Rondebosch, Cape Town
  - Newlands, Durban
  - Silverglen, Durban
  - Newtown, Johannesburg
  - Parktown, Johannesburg
  - Radiokop, Johannesburg
  - Stellenbosch, Western Cape
  - Cape Town
  - Durban
  - East London
  - Paarl
  - Pretoria
  - Soweto
  - Thabazimbi
  - Witbank
  - Worcester
- Spain (3):
  - A Coruña, Galicia
  - Barakaldo, Vizcaya
  - Mérida
- Lausanne, Switzerland
- Ukraine (6):
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Poltava
  - Vinnytsia

REFERENCES:
- [Derived] Topless R, Noorbaloochi S, Merriman TR, Singh JA. Change in serum urate level with urate-lowering therapy initiation associates in the immediate term with patient-reported outcomes in people with gout. Semin Arthritis Rheum. 2022 Oct;56:152057. doi: 10.1016/j.semarthrit.2022.152057. Epub 2022 Jun 29. PMID 35835008
- [Derived] Bardin T, Keenan RT, Khanna PP, Kopicko J, Fung M, Bhakta N, Adler S, Storgard C, Baumgartner S, So A. Lesinurad in combination with allopurinol: a randomised, double-blind, placebo-controlled study in patients with gout with inadequate response to standard of care (the multinational CLEAR 2 study). Ann Rheum Dis. 2017 May;76(5):811-820. doi: 10.1136/annrheumdis-2016-209213. Epub 2016 Nov 7. PMID 27821644
- See also: Related Info — http://www.gouttrial.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lesinurad 200 mg + Allopurinol: lesinurad 200 mg qd plus allopurinol
- Lesinurad 400 mg + Allopurinol: lesinurad 400 mg qd plus allopurinol
Period: Overall Study
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Started | 204 | 200 | 206
Completed | 163 | 150 | 158
Not Completed | 41 | 50 | 48
Not completed — Adverse Event | 4 | 12 | 9
Not completed — Gout flare | 3 | 0 | 2
Not completed — Protocol Violation | 8 | 15 | 12
Not completed — Sponsor terminated study | 5 | 2 | 3
Not completed — Lost to Follow-up | 5 | 7 | 11
Not completed — Withdrawal by Subject | 16 | 13 | 11
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol | Total
Number analyzed (Participants) | 204 | 200 | 206 | 610
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (11.1) | 51.3 (11.1) | 51.4 (10.6) | 51.2 (10.9)
Age, Customized [Number; unit: Participants]
  <65 | 184 | 175 | 185 | 544
  >=65 | 20 | 25 | 21 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 10 | 23
  Male | 197 | 194 | 196 | 587
Region of Enrollment [Number; unit: Participants]
  Australia | 4 | 9 | 4 | 17
  Belgium | 1 | 1 | 2 | 4
  Canada | 7 | 6 | 12 | 25
  Germany | 9 | 8 | 8 | 25
  New Zealand | 12 | 7 | 7 | 26
  Poland | 5 | 11 | 6 | 22
  South Africa | 30 | 36 | 33 | 99
  Spain | 2 | 4 | 2 | 8
  Switzerland | 1 | 0 | 0 | 1
  Ukraine | 25 | 24 | 25 | 74
  United States | 108 | 94 | 107 | 309

OUTCOME MEASURES:

1. Primary Outcome: Subjects With a Serum Urate (sUA) < 6.0 mg/dL by Month 6.
Description: Proportion of subjects with an sUA level that is < 6.0 mg/dL by Month 6.
Time Frame: 6 months
Population: Intent-to-Treat Population
Measure: Number; unit: Proportion of Subjects
Groups:
- Placebo + Allopurinol: placebo qd plus allopurinol
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 204 | 200 | 206
Proportion of Subjects | 0.554 | 0.665 | 0.233
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.32, 95% CI 2-sided [0.23 to 0.41], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.43, 95% CI 2-sided [0.34 to 0.52], Standard Error of Mean 0.05

2. Secondary Outcome: Gout Flares
Description: Mean rate of gout flares requiring treatment for the 6-month period from the end of Month 6 to the end of Month 12.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Gout Flares
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 204 | 200 | 206
Gout Flares | 0.7 (1.4) | 0.8 (1.7) | 0.9 (1.8)
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.5716, Negative Binomial Regression; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.57 to 1.37]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.7454, Negative Binomial Regression; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.60 to 1.45]

3. Secondary Outcome: Subjects With ≥ 1 Target Tophus at Baseline Who Experience Complete Resolution of at Least 1 Target Tophus by Month 12
Description: Proportion of subjects with ≥ 1 target tophus at Baseline who experience complete resolution of at least 1 target tophus by Month 12
Time Frame: 12 months
Measure: Number; unit: Proportion of Subjects
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Number analyzed (Participants) | 35 | 29 | 33
Proportion of Subjects | 0.314 | 0.276 | 0.333
Statistical Analysis 1: Comparison: Lesinurad 200 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.8466, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.02, 95% CI 2-sided [-0.24 to 0.2]
Statistical Analysis 2: Comparison: Lesinurad 400 mg + Allopurinol vs Placebo + Allopurinol; Test type: Superiority or Other; p = 0.6301, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.06, 95% CI 2-sided [-0.29 to 0.17]

ADVERSE EVENTS:
Arm/Group | Lesinurad 200 mg + Allopurinol | Lesinurad 400 mg + Allopurinol | Placebo + Allopurinol
Serious Adverse Events (participants affected / at risk) | 9/204 | 19/200 | 8/206
Other Adverse Events (participants affected / at risk) | 85/204 | 82/200 | 60/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Allopurinol (N=204) | Lesinurad 400 mg + Allopurinol (N=200) | Placebo + Allopurinol (N=206)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Allopurinol (N=204) | Lesinurad 400 mg + Allopurinol (N=200) | Placebo + Allopurinol (N=206)
Upper respiratory tract infection (Infections and infestations) | 14 (16) | 30 (39) | 21 (23)
Influenza (Infections and infestations) | 14 (17) | 8 (9) | 4 (4)
Bronchitis (Infections and infestations) | 9 (9) | 4 (4) | 4 (5)
Headache (Nervous system disorders) | 10 (11) | 12 (13) | 8 (8)
Hypertension (Vascular disorders) | 17 (17) | 16 (16) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 14 (21) | 7 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (24) | 6 (7) | 9 (14)
Blood creatinine increased (Investigations) | 8 (9) | 19 (24) | 7 (7)
Joint sprain (Injury, poisoning and procedural complications) | 9 (9) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.